CLINICAL TRIAL: NCT00994149
Title: Use for Diazoxide in the Initial Management of Hypoglycemia in Infants of Diabetic Mothers and Infants Large for Gestation
Brief Title: Diazoxide In the Management Of Hypoglycemic Neonates
Acronym: DIMOHN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Dr. Koravangattu Sankaran, University of Saskatchewan, Department of Pediatrics, Neonatal Research Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio-REB #08-151; HC Control Number: 126963
Record Dates: First submitted 2009-09-30; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Infant, Newborn, Diseases; Pregnancy in Diabetics; Infant, Diabetic Mother; Hypoglycemia; Infant, Large for Gestational Age
Keywords: Infants of Diabetic Mothers; Hypoglycemia; Diazoxide; Large for Gestation Infants
MeSH Terms: conditions — Infant, Newborn, Diseases; Pregnancy in Diabetics; Hypoglycemia | interventions — Diazoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diazoxide (Experimental): Infants in this are will receive 10mg/kg/d of diazoxide divided and given every eight hours
  Interventions: Drug: Diazoxide
- Ora-plus (Placebo Comparator): Liquid suspension modified to match intervention. Given every eight hours. Provided in shielded syringes.
  Interventions: Drug: Ora-plus

INTERVENTIONS:
Drug: Diazoxide — 10mg/kg/d divide every 8 hours
  Other Names: Brand Name: Proglycem
  Arms: Diazoxide
Drug: Ora-plus — placebo, give every 8 hours.
  Arms: Ora-plus

SUMMARY:
Diazoxide is an oral hyperglycemic medication. Diazoxide has been proven effective for treating hypoglycemia in infants and children with some types of persistent hyperinsulinemic hypoglycemia. The mechanism of action results in decreased insulin secretion. One of the causes of hypoglycemia in infants of diabetic mothers occurs due to a transient hyperinsulinemic state postnatally. The investigators have clinical experience and success using diazoxide in their unit for patients with hypoglycemia not adequately managed with intravenous (iv) dextrose and enteral supplementation. In this randomized controlled study the investigators expect that by using diazoxide as the initial treatment for infants of diabetic mothers with asymptomatic hypoglycemia (blood glucose of 2.5 to 2.0mmol/L), the investigators will be able to decrease the number of infants requiring an intravenous by at least thirty percent.

ELIGIBILITY:
Inclusion Criteria:

* Infants of diabetic mothers (IDMs) or infants weighing >90%
* Hypoglycemia: two consecutive blood glucose measurements <2.6mol/L and >1.9mmol/L in the first twelve hours of life
* > 36 weeks gestational age

Exclusion Criteria:

* Infants with symptomatic hypoglycemia (regardless of value
* Infants who meet criteria for intravenous dextrose according to the Canadian Pediatric Society (CPS) position statement
* Infants with contraindications for enteral feeds and/or medications

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Blood glucose measurement less than 2.0mmol/L | 14 days

SECONDARY OUTCOMES:
Number of infants with significantly low blood glucose measurements (<1.5mmol/L). | 14 days
Length of stay for infants in hospital | 14 days
Need for intravenous dextrose infusion to maintain blood glucose above 2.0mmol/L | 14 days
Admission to neonatal intensive care unit (NICU) | 14 days
Thrombocytopenia and/or Leukopenia | 14 days
Electrolyte imbalance requiring clinical intervention (intravenous or oral) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Koravangattu Sankaran, MD, BS, FRCPC, F.C.C.M., Principal Investigator — University of Saskatchewan, Department of Pediatrics, Head of Neonatal Research Group
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Screening guidelines for newborns at risk for low blood glucose. Paediatr Child Health. 2004 Dec;9(10):723-740. doi: 10.1093/pch/9.10.723. No abstract available. PMID 19688086
- [Background] Stenninger E, Flink R, Eriksson B, Sahlen C. Long-term neurological dysfunction and neonatal hypoglycaemia after diabetic pregnancy. Arch Dis Child Fetal Neonatal Ed. 1998 Nov;79(3):F174-9. doi: 10.1136/fn.79.3.f174. PMID 10194986
- [Background] Holtrop PC. The frequency of hypoglycemia in full-term large and small for gestational age newborns. Am J Perinatol. 1993 Mar;10(2):150-4. doi: 10.1055/s-2007-994649. PMID 8476480
- [Background] Cornblath M, Hawdon JM, Williams AF, Aynsley-Green A, Ward-Platt MP, Schwartz R, Kalhan SC. Controversies regarding definition of neonatal hypoglycemia: suggested operational thresholds. Pediatrics. 2000 May;105(5):1141-5. doi: 10.1542/peds.105.5.1141. PMID 10790476
- [Background] Diwakar KK, Sasidhar MV. Plasma glucose levels in term infants who are appropriate size for gestation and exclusively breast fed. Arch Dis Child Fetal Neonatal Ed. 2002 Jul;87(1):F46-8. doi: 10.1136/fn.87.1.f46. PMID 12091291
- [Background] Hoseth E, Joergensen A, Ebbesen F, Moeller M. Blood glucose levels in a population of healthy, breast fed, term infants of appropriate size for gestational age. Arch Dis Child Fetal Neonatal Ed. 2000 Sep;83(2):F117-9. doi: 10.1136/fn.83.2.f117. PMID 10952705
- [Background] Hawdon JM. Hypoglycaemia and the neonatal brain. Eur J Pediatr. 1999 Dec;158 Suppl 1:S9-S12. doi: 10.1007/pl00014319. PMID 10592092
- [Background] Stenninger E, Schollin J, Aman J. Early postnatal hypoglycaemia in newborn infants of diabetic mothers. Acta Paediatr. 1997 Dec;86(12):1374-6. doi: 10.1111/j.1651-2227.1997.tb14916.x. PMID 9475319
- [Background] Nold JL, Georgieff MK. Infants of diabetic mothers. Pediatr Clin North Am. 2004 Jun;51(3):619-37, viii. doi: 10.1016/j.pcl.2004.01.003. PMID 15157588
- [Background] DRASH A, WOLFF F. DRUG THERAPY IN LEUCINE-SENSITIVE HYPOGLYCEMIA. Metabolism. 1964 Jun;13:487-92. doi: 10.1016/0026-0495(64)90133-7. No abstract available. PMID 14193979
- [Background] Agrawal RK, Lui K, Gupta JM. Neonatal hypoglycaemia in infants of diabetic mothers. J Paediatr Child Health. 2000 Aug;36(4):354-6. doi: 10.1046/j.1440-1754.2000.00512.x. PMID 10940170
- [Background] Tyrrell VJ, Ambler GR, Yeow WH, Cowell CT, Silink M. Ten years' experience of persistent hyperinsulinaemic hypoglycaemia of infancy. J Paediatr Child Health. 2001 Oct;37(5):483-8. doi: 10.1046/j.1440-1754.2001.00748.x. PMID 11885714
- [Background] Touati G, Poggi-Travert F, Ogier de Baulny H, Rahier J, Brunelle F, Nihoul-Fekete C, Czernichow P, Saudubray JM. Long-term treatment of persistent hyperinsulinaemic hypoglycaemia of infancy with diazoxide: a retrospective review of 77 cases and analysis of efficacy-predicting criteria. Eur J Pediatr. 1998 Aug;157(8):628-33. doi: 10.1007/s004310050900. PMID 9727845
- [Background] Dunne MJ, Cosgrove KE, Shepherd RM, Aynsley-Green A, Lindley KJ. Hyperinsulinism in infancy: from basic science to clinical disease. Physiol Rev. 2004 Jan;84(1):239-75. doi: 10.1152/physrev.00022.2003. PMID 14715916
- [Background] Shirland L. When it is more than transient neonatal hypoglycemia: hyperinsulinemia--a case study challenge. Neonatal Netw. 2001 Jun;20(4):5-11. doi: 10.1891/0730-0832.20.4.5. PMID 12143902
- [Background] Taketomo CK, Hodding JH, Kraus DM. Pediatric Dosage Handbook 14th edition. Hudson (OH): Lexi-comp, Inc. 2007: 485-6
- [Background] McGraw ME, Price DA. Complications of diazoxide in the treatment of nesidioblastosis. Arch Dis Child. 1985 Jan;60(1):62-4. doi: 10.1136/adc.60.1.62. PMID 3970573
- [Background] Behrman RE, Kliegman R, Jenson HB, StantonBF. Nelson Textbook of Pediatrics 18th Edition. Philadelphia: WB Saunders Company 2007:783-6